CLINICAL TRIAL: NCT03365596
Title: Functional MRI and DTI Study for Brain Network Analysis and Recovery Prediction in Subacute Stroke Patients
Brief Title: Recovery Prediction of Motor Function Using Neuroimaging Techniques in Subacute Stroke Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02-107
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2019-07

CONDITIONS: Stroke
Keywords: Brain connectivity; Magnetic resonance imaging; Recovery prediction
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subacute stroke
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Conventional therapy — According to the status of a patient, optimized therapy will be applied.

SUMMARY:
Prediction of recovery from stroke can assist in the planning of impairment-focused rehabilitation. To achieve better prediction for clinical purposes, this study investigated a new prediction model with low inter-individual variability and high accuracy using neuroimaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke patients
* Unilateral stroke
* Subacute stage (less than 4 weeks)

Exclusion Criteria:

* Major active neurological disease or psychiatric disease
* A history of seizure
* Metallic implants in their brain

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-ever stroke patients at subacute stage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment score at 3 months after stroke onset | 3 months after stroke onset
  Measurement of motor function of upper and lower extremities

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No